CLINICAL TRIAL: NCT00464607
Title: A Prospective, Randomized, Controlled Clinical Study on the Assessment of Tolerability and of Clinical Efficacy of MERIONAL® (hMG-IBSA) Administered Subcutaneously Versus MERIONALâ Administered Intramuscularly in Women Undergoing Controlled Ovarian Hyperstimulation (COH) in an ART Programme (IVF)
Brief Title: Prospective, Randomized, Controlled, Clinical Study on Tolerability and Efficacy of hMG-IBSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00IF/HMG06
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2007-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — hMG-IBSA; Ovulation Induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: hMG-IBSA
Procedure: Ovarian stimulation

SUMMARY:
Purpose of the study is the evaluation of the tolerability (both local and systemic) and the clinical efficacy (in terms oocytes recovered) of subcutaneously versus intramuscularly administered Merional® (IBSA, Lugano - CH) in patients undergoing controlled ovarian hyperstimulation (COH) in an ART programme (IVF).

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* aged between 20 and 40 years
* undergoing ovarian stimulation for the purposes of oocyte retrieval in an assisted conception programme
* Body Mass Index (BMI) 20-28 kg/m2
* early follicular phase FSH level < 9 IU/l.

Exclusion Criteria:

* ascertained or presumptive hypersensitivity to the active principle and/or their ingredients
* primary ovarian failure
* ovarian cysts or enlargement not due to polycystic ovarian syndrome
* oocyte donation
* abnormal bleeding of undetermined origin
* patients who have exhibited poor response or requiring doses of more than 300 IU daily in previous treatment cycles or those who have received similar therapies (previous treatment cycles) in the 30 days prior to the beginning of the present study
* uncontrolled thyroid or adrenal dysfunction
* neoplasia
* severe impairment of the renal and/or hepatic functions
* diabetes and active thrombophlebitis, cardiopathies and epilepsy
* presence of clinically significant systemic disease or any contraindication of being pregnant and/or carrying out a pregnancy to term
* presence of any anatomical abnormality of the reproductive system
* being pregnant or breastfeeding
* menopause

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160
Dates: Start 2001-12; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Number of oocytes recovered

SECONDARY OUTCOMES:
Efficacy: Day of Oocyte collection, 17β-estradiol Cmax, Total dose of gonadotrophin (IU) or n° of vials and n° of vials/day,Number of mature follicles (follicles ³ 16 mm in diameter) on hCG day (or one day earlier), Clinical pregnancy rate
Tolerability: Number of Adverse Events (AEs) experienced during the study, Occurrence of Ovarian Hypestimulation Syndrome (OHSS), Local tolerability at the injection site, Haematological-biochemical laboratory tests, before and after treatment,

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Ragni, Prof., Principal Investigator — Ospedale S.Martino - Genova (Italy); Luigi Fedele, Prof., Principal Investigator — Ospedale S. Paolo - Milano (Italy); Giuseppe De Placido, Prof., Principal Investigator — Ospedale Federico II - Napoli (Italy); Marco Massobrio, Prof., Principal Investigator — Ospedale S. Anna - Torino (Italy)
Locations (4):
- Italy (4):
  - Ospedale S. Martino, Genova, Genova
  - Ospedale S. Paolo, Milan, Milano
  - Ospedale Federico II, Napoli, Napoli
  - Ospedale S. Anna, Torino, Torino